CLINICAL TRIAL: NCT04423406
Title: The Changes in Carotid Plaque Neovascularization After Long-term Elovocumab Injection Therapy: A Follow-Up Study by Contrast Enhanced Ultrasonography
Brief Title: The Changes in Carotid Plaque Neovascularization After Elovocumab Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zibo Central Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZiboCH1
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
150 selected patients will be recruited, who have at least one atherosclerotic plaque in the carotid artery that is thicker than 2.0 mm and which is determined to be uniformly or predominantly echolucent by standard ultrasonography. For each of the plaques, standard ultrasonography will be used to evaluate lesion echogenicity, while contrast-enhanced ultrasonography (CEUS) will be used to perform the visual and quantitative analysis of neovascularization. Each technique will be applied at baseline (at the time of study enrollment) and following 0.5、1 year of Elococumab Injection treatment. During the study, these patients will be treated with Elococumab Injection (1ml:140mg),ih, every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. have at least one atherosclerotic plaque in the carotid artery that is thicker than 2.0 mm and which is determined to be uniformly or predominantly echolucent by standard ultrasonography;
* 2.patients were referred for optimal medical treatment;
* 3.patients agreed to undergo follow-up CEUS at half-year and 1-year interval.

Exclusion Criteria:

* 1.patients had previous history of cerebral thrombosis or cerebral embolism;
* 2.patients were contraindicated to the usage of contrast media;
* 3.image quality of baseline or follow-up CEUS was severely impaired (in presence of severe artifact, non-diagnostic);
* 4.patients withdrew the informed consents during follow-up;
* 5.patients experienced major adverse cerebrovascular events during follow-up;
* 6.patients refused to undergo follow-up CEUS;
* 7.lost follow-up

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 150 eligible coronary atherosclerosis disease patients were anticipated to include in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-27 (Estimated)

PRIMARY OUTCOMES:
The Changes in Carotid Plaque Neovascularization | June 2020 to December 2021
  We will use the time-signal intensity curve to calculate the changes in carotid plaque neovascularization.The time-intensity curve parameters includes: Baseline intensity(BI) and peak intensity (PI).Due to the ultrasound contrast agent, the intra-plaque signal intensity increased. Thus, enhanced intensity (EI) was calculated as follows: EI = PI - BI. EI is a parameter that measures the intensity differences between pre- and post-injections of the intravascular tracer. Relative plaque enhancement (EI-R), measured at the separate peak enhancement point in the blood and plaque, will be calculated as the ratio of enhanced intensity in the carotid artery lumen (EI-L) to the enhanced intensity in the plaque (EI-P) using the following formula: EI-R=EI-L/EI-P.

OTHER OUTCOMES:
The Changes in Carotid Plaque Size | June 2020 to December 2021
  After one year's treatment of Elovocumab Injection, the patients will undergo follow-up standard ultrasonography again. We will measure the size of each lesion.The carotid plaque sizes at pre- and post-elovocumab therapy will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Li, Principal Investigator — Zibo Central Hospital
Locations (1):
- Zibo Central Hospital, Zibo, Shandong, China

REFERENCES:
- [Derived] Chen J, Zhao F, Lei C, Qi T, Xue X, Meng Y, Zhang W, Zhang H, Wang J, Zhu H, Cheng C, Wang Q, Bi C, Song B, Jin C, Niu Q, An F, Li B, Huo X, Zhao Y, Li B. Effect of evolocumab on the progression of intraplaque neovascularization of the carotid based on contrast-enhanced ultrasonography (EPIC study): A prospective single-arm, open-label study. Front Pharmacol. 2023 Jan 4;13:999224. doi: 10.3389/fphar.2022.999224. eCollection 2022. PMID 36686711